CLINICAL TRIAL: NCT04728399
Title: Effects of Soy Peptide and Conjugated Linoleic Acid on Body Composition: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Soy Peptide, Conjugated Linoleic Acid, Overweight or Obese, Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fangfang Zeng (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Fangfang Zeng, Associate Professor, School of basic medicine and public health, Jinan University Guangzhou
Organization: Jinan University Guangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JNUKY-2020-002
Record Dates: First submitted 2021-01-15; First posted 2021-01-28 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Overweight or Obesity
Keywords: Soy Peptide; Conjugated Linoleic Acid; Overweight or Obesity; Body Composition; Fatty liver disease; RCT
MeSH Terms: conditions — Overweight; Obesity; Non-alcoholic Fatty Liver Disease | interventions — Control Groups; Proteins; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 2g Soybean peptide, 3g CLA and ng protein.
  Interventions: Dietary Supplement: Experimental group
- Control group (Placebo Comparator): 2g+N protein and 3g Soybean oil.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Experimental group — Take 1 bag a day with warm boiling water. Intervention: 2g Soybean peptide, 3g CLA and ng protein. They will complete all baseline, 12-weeks, and 24-weeks visits
  Other Names: Soybean peptide and CLA
  Arms: Experimental group
Dietary Supplement: Control group — Take 1 bag a day with warm boiling water. Intervention: 2g+N protein and 3g Soybean oil. They will complete all baseline, 12-weeks, and 24-weeks visits
  Other Names: Protein and Soybean oil
  Arms: Control group

SUMMARY:
Soybean peptides are a mixture of active peptides obtained from the hydrolysis of soybean protein, which have biological activities such as antioxidant, blood pressure lowering, anti-fatigue and lipid lowering, etc. They can regulate food intake, increase satiety, and reduce fat body ratio by reducing cholesterol and triglyceride content and stimulating CCK secretion.Conjugated linoleic acid (CLA) is a set of linoleic acid with conjugated unsaturated double bond, the location and structure of the isomers have been approved by the ministry of health in China as a new resource food , widely used in areas such as health care products, functional foods and food additives, animal experiments showed that it has reduce tumor, atherosclerosis, obesity risk.Therefore, in this study, the effect of conjugated linoleic acid combined with soybean peptide on overweight and obese people was investigated in a randomized controlled manner.

DETAILED DESCRIPTION:
Aim 1: To test the effects of combined supplementation of soybean peptide and conjugated linoleic acid on body fat, liver fat and muscle content of overweight and obese people;Aim 2: To test the effects of combined supplementation of soybean peptide and conjugated linoleic acid on blood lipid, blood glucose, fat or inflammatory factors in overweight and obese people; Aim 3: Test the impact of the above interventions on safety indicators (safety indicators: liver and kidney function, self-reported adverse reactions or diseases). Aim 4: To provide scientific basis for the development of functional food for weight loss and muscle gain.The public health significance of this research is that find a new functional food for weight loss and muscle gain.

ELIGIBILITY:
Inclusion Criteria:

* Age - 18-65 years old;
* Gender-not limited;
* BMI-24-35 kg/m2;
* Body fat rate-Male ≥25%, female ≥30% (body fat meter can be used for screening, DXA is used for diagnosis);
* Waist circumference: male >90cm, Female>80cm (not required).

Exclusion Criteria:

* Suffer from serious diseases such as heart, liver, kidney, brain, hematopoietic, immune, thyroid, malignant tumors;
* Take drugs or supplements that have a known effect on body fat and muscle mass;
* Those whose weight has changed more than 10% in the past 3 months;
* Those who have cognitive or mental disorders and cannot conduct questionnaire surveys;
* People who are physically disabled and cannot walk normally;
* Those whose compliance with the pre-experiment period cannot meet the requirements;
* Fail to sign the informed consent form, or other researchers think it is not suitable for participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | Baseline & 24weeks
  Liver fat content will be measured by magnetic resonance (MR) which will be evaluated for change over the course of liver fat content.
  Baseline: Evaluate the initial fat content of the subjects; 24weeks: Evaluate whether the fat content of the subjects changes after the intervention.
Fat and thin tissue | Baseline & 12 weeks & 24weeks
  Body fat percentage will be screened with DXA apparatus.Assess the patient's physical condition.
  Baseline: Evaluate the body composition of the subjects to see whether they meet the inclusion criteria; 12 weeks: After 3 months of intervention, If the percentage of fat is lower than the baseline, the body composition is improved, if the proportion of fat increased by more than 5%, the test should be stopped in time.
  24 weeks: Evaluate the improvement of body composition before and after the intervention. If the percentage of fat is lower than the baseline, the body composition is improved.
  Baseline: Evaluate the body composition of the subjects to see whether they meet the inclusion criteria; 12 weeks: After 3 months of intervention, the subjects will be evaluated for weight improvement.If the proportion of fat; 24 weeks: Evaluate the improvement of body composition before and after the intervention.
Adipocytokine | Baseline & 24weeks
  Adipocytokines will be detected by biochemical experiments to reveal the possible pathways of action of soybean peptides and conjugated linoleic acid.
  Baseline: Evaluate the levels of adipocytokines (such as leptin and adiponectin) before intervention; 24 weeks: Evaluate the levels of adipocytokines (such as leptin and adiponectin) after intervention, If the serum leptin and adiponectin levels change, it can provide a new idea for the combined weight loss mechanism of soybean peptide and conjugated linoleic acid.
Inflammatory factor index | Baseline & 24weeks
  Inflammatory factor index will be detected by biochemical experiments to reveal the possible pathways of action of soybean peptides and conjugated linoleic acid.
  Baseline: Evaluate the levels of inflammatory factors (such CRP, IL-6) before intervention; 24weeks: Evaluate the levels of inflammatory factors after intervention, If the levels of inflammatory factors change, it suggests that soy peptides and conjugated acid oil may achieve weight loss through inflammatory pathway.
Blood fat | Baseline & 12 weeks & 24weeks
  Blood fat inde(such as TG, TC) will be detected by biochemical examination. Baseline: assess the physical condition of subjects to determine whether they meet the criteria for inclusion; 12 weeks: Evaluate the levels of TG, TC after three-months intervention, If there is a significant increase in Blood fat, the experiment should be stopped in time; 24 weeks: Evaluate the effect of lowering blood lipid of the subjects.

SECONDARY OUTCOMES:
Liver function | Baseline & 12 weeks & 24weeks
  Liver function(such as AST, ALT) will be detected by biochemical examination.It is safety index to assess physical condition.
  Baseline: Assess whether the liver function of the subjects is normal; 12 weeks: After 3 months intervation, assess the change in liver function, If the liver function is damaged, the experiment should be terminated in time.
  24 weeks: After intervation, assess the change in liver function.
Food recording | Baseline & 12 weeks & 24weeks
  3-d dietary records will be used for food recording. Used to assess the subjects' other energy intake. The heading includes food type, cooking style and consumption amount.
Wechat steps | Baseline & 12 weeks & 24weeks
  Record the 3-day wechat steps in kilograms to assess basic movement situation.
Sitting time | Baseline & 12 weeks & 24weeks
  Record the 3-day sitting time in hours to evaluate the sedentary situation of subjects every day.
Regular sport recording | Baseline & 12 weeks & 24weeks
  Record the 3-day regular movement, including the name and duration of movements on that day.（e.g., swimming, two hours）
Kidney function | Baseline & 12 weeks & 24weeks
  Kidney function(such as Urea, creatinine) will be detected by biochemical examination.It is safety index to assess physical condition.
  Baseline: Assess whether the kidney function of the subjects is normal; 12 weeks: After 3 months intervation, assess the change in kidney function, If the kidney function is damaged, the experiment should be terminated in time.
  24 weeks: After intervation, assess the change in kidney function.

OTHER OUTCOMES:
Anxiety situation | Baseline & 12 weeks & 24weeks
  SAS scale will be used to reflect the subject's mood.Generally speaking, the total score of anxiety is less than 50 points for normal;50 to 60 people have mild anxiety, 61 to 70 people have moderate anxiety, and 70 or more people have severe anxiety.
Adverse reactions or side effects | Baseline & 12 weeks & 24weeks
  ) Patients were questioned by investigators at baseline, 12 weeks and 24 weeks respectively. If there is any suspicious incident, it will be reported by the investigator first, and then reviewed by the doctor or the project leader and recorded in time.
Compliance assessment | 12 weeks & 24weeks
  Compliance was assessed at week 12 and 14 using the MMAS-8 questionnaire. There are 8 items in total. For questions 1-4 and 6-7, if you choose "no", you will get 1 point; for question 5, if you choose "yes", you will get 1 point; for other options, you will get 0 point; for question 8, if you choose "never, rarely, sometimes, often", you will get 1 point, 0.75 point, 0.5 point, 0.25 point and 0 point respectively. Less than 6 points indicated poor compliance, 6-8 points indicated medium compliance, and 8 points indicated good compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Derakhshande-Rishehri SM, Mansourian M, Kelishadi R, Heidari-Beni M. Association of foods enriched in conjugated linoleic acid (CLA) and CLA supplements with lipid profile in human studies: a systematic review and meta-analysis. Public Health Nutr. 2015 Aug;18(11):2041-54. doi: 10.1017/S1368980014002262. Epub 2014 Nov 7. PMID 25379623
- [Result] Bruen R, Fitzsimons S, Belton O. Atheroprotective effects of conjugated linoleic acid. Br J Clin Pharmacol. 2017 Jan;83(1):46-53. doi: 10.1111/bcp.12948. Epub 2016 May 7. PMID 27037767
- [Result] den Hartigh LJ. Conjugated Linoleic Acid Effects on Cancer, Obesity, and Atherosclerosis: A Review of Pre-Clinical and Human Trials with Current Perspectives. Nutrients. 2019 Feb 11;11(2):370. doi: 10.3390/nu11020370. PMID 30754681
- [Result] Whigham LD, Watras AC, Schoeller DA. Efficacy of conjugated linoleic acid for reducing fat mass: a meta-analysis in humans. Am J Clin Nutr. 2007 May;85(5):1203-11. doi: 10.1093/ajcn/85.5.1203. PMID 17490954
- [Result] Fuke G, Nornberg JL. Systematic evaluation on the effectiveness of conjugated linoleic acid in human health. Crit Rev Food Sci Nutr. 2017 Jan 2;57(1):1-7. doi: 10.1080/10408398.2012.716800. PMID 27636835